CLINICAL TRIAL: NCT04678011
Title: A Personalized Surveillance and Intervention Protocol for Patients With Familial Adenomatous Polyposis That Have Undergone (Procto)Colectomy
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Leiden University Medical Center (Other); The Netherlands Cancer Institute (Other); St Mark's Hospital Foundation (Other); Hospital Clinic of Barcelona (Other); Hôpital Edouard Herriot (Other); Maria Sklodowska-Curie National Research Institute of Oncology (Other); Hospital General Universitario de Alicante (Other); University Medical Center Mainz (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Prof. Evelien Dekker, MD, PhD, Prof. dr. Evelien Dekker, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W20_182
Record Dates: First submitted 2020-11-24; First posted 2020-12-21 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Familial Adenomatous Polyposis
Keywords: Endoscopic surveillance; Endoscopic interventions; Personalised care; Gastrointestinal neoplasia
MeSH Terms: conditions — Adenomatous Polyposis Coli

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Personalized surveillance and intervention protocol
  Interventions: Procedure: Personalized surveillance and intervention protocol

INTERVENTIONS:
Procedure: Personalized surveillance and intervention protocol — This study uses one arm. Participants will undergo endoscopic surveillance with intervals between 6 months and 2 years, depending on severity of polyposis and performed endoscopic interventions.

SUMMARY:
The purpose of this study is to determine the efficacy and safety of a personalised surveillance and intervention protocol for patients with familial adenomatous polyposis (FAP) that have undergone (procto)colectomy.

DETAILED DESCRIPTION:
Familial adenomatous polyposis (FAP) is characterized by formation of up to hundreds to thousands of polyps throughout the entire colon and rectum. When left untreated, nearly all patients with FAP develop colorectal cancer at a median age of 35-45 years. To prevent colorectal cancer in patients with FAP, prophylactic colorectal surgery is performed. The preferred surgical procedures for FAP are a restorative proctocolectomy with ileal pouch-anal anastomosis (IPAA) or a subtotal colectomy with ileorectal anastomosis (IRA) or ileosigmoidal anastomosis (ISA).

After both types of prophylactic colorectal surgery, subtotal colectomy with IRA/ISA or proctocolectomy with IPAA, patients will require life-long surveillance because disease progression and development of new adenomas in retained rectum, pouch or residual rectal cuff will occur.

The 10-years risk of developing one or more adenomas in the rectum after IRA is 100% compared to 33% in the pouch after IPAA. The risk of developing rectal cancer after IRA was found to be 9% and 11% in two large studies with a median follow-up of 12.8 and 15 years, respectively. One study showed that the 10-years risk of developing a carcinoma in the pouch was 1%. As patients are usually operated at a young age, and nowadays have a long life-expectancy, the actual cumulative life-time risk will presumably be higher.

The recently published ESGE (European Society of Gastrointestinal Endoscopy) polyposis guideline recommends a one to two yearly endoscopic surveillance interval after prophylactic colorectal surgery in FAP, both for patients that underwent IRA/ISA and IPAA, with removal of all polyps >5mm. This recommendation is based on expert-opinion, since no studies have been reported comparing the efficacy and safety of different surveillance intervals. No advices are provided on which patients will benefit from which surveillance interval.

With the proposed study, the investigators aim to provide evidence for personalized endoscopic surveillance for patients with FAP that have undergone (procto)colectomy with construction of an IRA/ISA or IPAA with the goal to prevent development of advanced neoplasia (AN) by endoscopically removing lesions before they progress to AN.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of FAP, at least one of following: genetic diagnosis (proven APC germline mutation) and/or clinical diagnosis (>100 colorectal adenomas in combination with a positive family history of FAP)
* Have undergone prophylactic (procto)colectomy with IRA/ISA or IPAA
* Age 18 years or older

Exclusion Criteria:

* Not able to remove all polyps with an indication for removal during (multiple) clearing endoscopies
* Cancer at baseline endoscopy
* Need for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with FAP treated at one of the participating centres.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-11-24 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Advanced neoplasia | Up to 5 years
  Incidence of advanced neoplasia (advanced adenoma and cancer). An advanced adenoma is defined as size ≥ 10mm and/or high-grade dysplasia. This surveillance and intervention protocol will be considered successful when the incidence of advanced neoplasia is less than 5% after a study period of 5 years.

SECONDARY OUTCOMES:
Characteristics polyps | Up to 5 years
  Incidence and characteristics of polyps detected/removed in patients with IRA/ISA and IPAA
Radicality of different endoscopic intervention techniques | Up to 5 years
  Rate of radical endoscopic interventions
Feasibility endoscopic interventions | Up to 5 years
  Incidence of lesions not amenable to endoscopic removal
Surgical interventions | Up to 5 years
  Incidence of surgical interventions
Surveillance burden | Up to 5 years
  Surveillance burden (number of endoscopies per patient)
Complications | Up to 5 years
  Incidence of endoscopy related complications

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Centre, Amsterdam, North Holland, Netherlands